CLINICAL TRIAL: NCT01147185
Title: Effectiveness of Automated Locomotor Training in Patients With Acute Incomplete Spinal Cord Injury: A Multicenter Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMSCI-DR
Record Dates: First submitted 2010-05-07; First posted 2010-06-22 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injuries, Locomotor training, Dose-Response
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive training (Other): Locomotor training using a robotic device of at least 50 minutes
  Interventions: Device: Locomotor training using a robotic device
- Standard training (Active Comparator): Locomotor training using a robotic device of maximally 25 minutes
  Interventions: Device: Locomotor training using a robotic device

INTERVENTIONS:
Device: Locomotor training using a robotic device — 50min walking time, 3-5 trainings/week.
  Other Names: Lokomat, Hocoma AG, Volketswil/Switzerland
  Arms: Intensive training
Device: Locomotor training using a robotic device — 25min walking time, 3-5 trainings/week.
  Other Names: Lokomat, Hocoma AG, Volketswil/Switzerland
  Arms: Standard training

SUMMARY:
The purpose of this study is to determine whether longer locomotor training results in a mor favorable outcome in patients with incomplete spinal cord injury.

DETAILED DESCRIPTION:
About half of patients who experience a traumatic spinal cord injury (SCI) have still motor and/or sensory function below the level of the lesion. A large proportion of these patients become ambulatory within the first six months after the SCI. In order to optimally train the walking function patients are partially unloaded from their body weight while they walk on a moving treadmill. In severe cases therapists have to assist the leg movements which is an exhaustive work limiting training time. In the last few years robotic devices have been developed which enable longer training time. Studies evaluating the training of patients with hemiparesis showed that longer training time is associated with a better outcome. The present study aims at evaluating the effect of training time within the robotic device on the recovery of ambulatory function. Subject with an acute incomplete SCI will be included. The intervention consist of a walking training which lasts at least 50min, the training of the control group last at maximum 25min. Both groups will undergo 3-5 trainings per week. Group assignment will be performed at random. The study lasts for 8 weeks. The primary outcome will be the self selected walking speed which will be assessed bi-weekly during the training period and 4 months later.

ELIGIBILITY:
Inclusion Criteria:

* patients with spinal cord injury (SCI) categorized according to the standard classification of the American Spinal Injury Association as ASIA B or C within the first two weeks after trauma
* traumatic etiology of SCI
* limited walking ability (Walking Index for Spinal Cord Injury ≤5)
* able to start training or rehab within 60 days after trauma
* motor level between cervical 4 and thoracic 12
* signed informed consent

Exclusion Criteria:

* exclusion criteria of the Lokomat:(bodyweight > 130kg, body height > 200cm, leg length diff > 2cm, osteoporosis, instable fracture of lower extremity, restricted range of motion, decubitus ulcer of lower extremity)
* concomitant injury limiting walking ability (e.g. lower extremity fractures, instable spine fractures, Joint instability preventing weight-bearing, severe soft tissue lesion)
* pre-existing medical conditions interfering with unrestricted walking (e.g. total joint replacement, pain, osteoarthritis, polyneuropathy, cardiopulmonary disease)
* age older than 65 years or younger than 18 years
* conus medullaris or cauda equina syndrome
* traumatic brain injury
* passive range of motion of the hips, knees and ankles not sufficient to allow normal kinematics consistent with upright gait
* patient participates in other rehabilitation or pharmacological study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Ten meter walking test | at start of training, at weeks 2, 4, 6, 8, 6 and 24
  Self selected walking speed over a distance of 10m

SECONDARY OUTCOMES:
Walking Index for Spinal Cord Injury (WISCI) | at start of training, at weeks 2, 4, 6, 8, 6 and 24
  Classification of walking ability on a rank ordered scale with 21 categories.
Spasticity | at start of training, at weeks 2, 4, 6, 8, 6 and 24
  Muscle tone is rated using the modified Ashworth and the Pess spasm frequency tests
Perceived exertion | after every training
Spinal Cord Independence Measure | at start of training, at weeks 2, 4, 6, 8, 6 and 24
Spinal cord injury classification | at start of training, at weeks 2, 4, 6, 8, 6 and 24
  Classification according to the standards by the American Spinal Cord Injury Association (ASIA)
Patients' Global Impression of Change Scale | At week 8

CONTACTS AND LOCATIONS:
Overall Officials: Markus Wirz, PT PhD, Principal Investigator — Zurich University of Applied Sciences
Locations (4):
- Berufsgenossenschaftliche Unfallklinik Murnau, Murnau am Staffelsee, Germany
- Spain (2):
  - Institut Guttmann, Barcelona
  - Hospital Nacional de Parapléjicos, Toledo
- Balgrist University Hospital, Zurich, Switzerland

REFERENCES:
- [Derived] Wirz M, Bastiaenen C, de Bie R, Dietz V. Effectiveness of automated locomotor training in patients with acute incomplete spinal cord injury: a randomized controlled multicenter trial. BMC Neurol. 2011 May 27;11:60. doi: 10.1186/1471-2377-11-60. PMID 21619574